CLINICAL TRIAL: NCT01805050
Title: Arthroscopically Repair of the Anterior Instability of the Shoulder Due an HAGL - Lesion - A Case Serie
Brief Title: Case Study: HAGL-lesion (HAGL:Humeral Avulsion Glenohumeral Ligament)
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Matthias Flury, Principal Investigator (Department of Upper Extremity), Schulthess Klinik
Other Study IDs: HAGL
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Shoulder Injuries and Disorders
Keywords: HAGL; Shoulder instability
MeSH Terms: conditions — Shoulder Injuries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- New Technique: All patients who underwent surgical repair of the anterior instability due an HAGL lesion.
  Interventions: Procedure: Arthroscopically repair of the anterior shoulder instability

INTERVENTIONS:
Procedure: Arthroscopically repair of the anterior shoulder instability — Arthroscopically repair of the anterior shoulder instability

SUMMARY:
This study shows a new technique which has been implemented at the schulthess clinic to improve the outcome after an correction of an anterior instability in the shoulder joint due to a HAGL lesion.

DETAILED DESCRIPTION:
The aim of the study is to describe and document the results of a case serie after an arthroscopically intervention to correct the anterior instability in the shoulder joint with one primary parameter (WOSI-Score) and several secondary parameters, which are used in the daily clinical routine (e.g.clinical examination, several questionnaires). The results of these parameters will be used to document the mid-term results (> 1 year after surgery).

ELIGIBILITY:
Inclusion Criteria:

* arthroscopically repair of the anterior instability of the shoulder due an HAGL lesion (performed by Dr. M. Flury, Dr. H.-K. Schwyzer or Dr. Ph. Frey at the Schulthess Klinik)
* patients ≥18 years
* written informed consent

Exclusion Criteria:

* additional surgeries at the affected side after the index surgery (arthroscopically repair of the anterior instability due an HAGL lesion)
* non-compliance
* disorders which handicap or inhibit the patient to follow the orders of the clinical testers
* request of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent surgical repair of the anterior instability due an HAGL lesion at the Schulthess Klinik and have been performed surgery by Dr. M. Flury, Dr. H.-K. Schwyzer or Dr. Ph. Frey
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
WOSI-Score | expected average of 2 years

SECONDARY OUTCOMES:
Sociodemographic Dates | expected average of 2 years
x-ray images | expected average of 2 years
Constant-Murley Score | expected average of 2 years
Rowe - Score | expected average of 2 years
SSV (Simple Shoulder Value) | expected average of 2 years
SST (Simple Shoulder Test) | expected average of 2 years
Measurement of the abduction strength | expected average of 2 years
Measurement of the external rotation strength | expected average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Flury, Dr, Principal Investigator — Upper Extremities Department
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zürich, Switzerland